CLINICAL TRIAL: NCT06457997
Title: First-in-Human, Phase 1b Study of PHN-010, an Antibody Drug Conjugate, in Patients With Advanced Solid Tumors
Brief Title: A Study of PHN-010 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated by Sponsor for strategic reasons.
Sponsor: Pheon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PHN-010-001
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Colon Cancer; Endometrial Cancer; Ovarian Cancer; Cervical Cancer; Advanced Solid Tumor; Advanced Cancer
Keywords: Antibody-Drug Conjugate; Carcinoma; Cancer; Solid Tumor
MeSH Terms: conditions — Lung Neoplasms; Colonic Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Carcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1a and Phase 1b (Experimental): PHN-010 is administered intravenously.
  Interventions: Drug: PHN-010

INTERVENTIONS:
Drug: PHN-010 — PHN-010 is an ADC

SUMMARY:
This first-in-human study will evaluate safety, tolerability, anti-tumor activity, immunogenicity, pharmacokinetics and pharmacodynamics of PHN-010, a novel antibody-drug conjugate (ADC), in patients with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Has histologically confirmed, advanced/metastatic:

  1. Colorectal adenocarcinoma (CRC), or
  2. Serous, endometroid, or clear-cell epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer, or
  3. Serous, endometroid or clear-cell endometrial cancer, or
  4. Adenocarcinoma or squamous-cell carcinoma of the cervix, or
  5. Non-small cell lung cancer (NSCLC).
* Has received at least one prior systemic therapy and radiologically or clinically determined progressive disease during or after the most recent line of therapy, and for whom no further standard therapy is available or who is intolerant to standard therapy.
* Has measurable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has adequate organ function.
* Has available tumor tissue sample at screening (either an archival specimen collected ≤ 3 years prior to the date of informed consent or fresh biopsy material).

Exclusion Criteria:

* Had prior treatment with any ADC containing topoisomerase-1 inhibiting payload.
* Has unstable central nervous system metastasis.
* Has persistent toxicities from previous systemic anti-cancer treatments of Grade >1.
* Has received systemic anti-neoplastic therapy within five half-lives or 21 days, whichever is shorter, prior to first dose of the study drug.
* Has received wide-field radiotherapy (> 30% of marrow-bearing bones) within 28 days, or focal radiation for analgesic purpose or for lytic lesions at risk of fracture within 14 days prior to first dose of the study drug, or no recovery from side effects of such intervention.
* Had major surgery (not including placement of vascular access device or tumor biopsies) within 28 days prior to first dose of the study drug, or no recovery from side effects of such intervention.
* Has acute and/or clinically significant bacterial, fungal, or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV).
* Has a history of non-infectious pneumonitis (NIP) / interstitial lung disease (ILD) requiring systemic steroids, active NIP / ILD or suspected NIP / ILD which cannot be ruled out by imaging for Screening.

Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (Phase 1a) | 18 months
Type, incidence and severity of adverse events (AEs) and serious adverse events (SAEs) (Phase 1a) | 18 months
Frequency of dose interruptions, reductions, and discontinuations (Phase 1a and 1b) | 18 months
Overall response rate (ORR) (Phase 1b) | 36 months

SECONDARY OUTCOMES:
Best overall response (BOR) (Phase 1a and 1b) | 36 months
Disease control rate (DCR) (Phase 1a and 1b) | 36 months
Progression free survival (PFS) (Phase 1a and 1b) | 36 months
Time to response (TTR) (Phase 1a and 1b) | 36 months
Overall survival (OS) (Phase 1a and 1b) | 36 months
Cancer antigen 125 (CA-125) response (Phase 1a and 1b) | 36 months
Time to CA-125 response (Phase 1a and 1b) | 36 months
Pharmacokinetics, maximum concentration (Cmax) of total ADC (Phase 1a and 1b) | 36 months
Pharmacokinetics, Cmax of total antibody (Phase 1a and 1b) | 36 months
Pharmacokinetics, Cmax of free payload (Phase 1a and 1b) | 36 months
Pharmacokinetics, time of Cmax (Tmax) of total ADC (Phase 1a and 1b) | 36 months
Pharmacokinetics, Tmax of total antibody (Phase 1a and 1b) | 36 months
Pharmacokinetics, Tmax of free payload (Phase 1a and 1b) | 36 months
Pharmacokinetics, area under the curve (AUC) of total ADC (Phase 1a and 1b) | 36 months
Pharmacokinetics, AUC of total antibody (Phase 1a and 1b) | 36 months
Pharmacokinetics, AUC of total free payload (Phase 1a and 1b) | 36 months
Pharmacokinetics, terminal half-life (t1/2) of total ADC (Phase 1a and 1b) | 36 months
Pharmacokinetics, t1/2 of total antibody (Phase 1a and 1b) | 36 months
Pharmacokinetics, t1/2 of free payload (Phase 1a and 1b) | 36 months
Concentration of anti-drug antibodies (Phase 1a and 1b) | 36 months
Type, incidence and severity of AEs and SAEs (Phase 1b) | 18 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - AdventHealth, Orlando, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT - San Antonio, San Antonio, Texas
  - NEXT - Virginia, Fairfax, Virginia
  - University of Washington/Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No